CLINICAL TRIAL: NCT05486026
Title: Efficacy of Duloxetine Compared to NSIADs in Osteoarthritis of Knee: A Randomized Open Labelled Clinical Trial
Brief Title: Efficacy of Duloxetine Compared to NSIADs in Osteoarthritis of Knee
Acronym: Duloxetine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Aryan Mohamadfatih Jalal, principal investigator, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Efficacy of Duloxetine
Record Dates: First submitted 2022-07-31; First posted 2022-08-03 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-11

CONDITIONS: Osteo Arthritis Knee
Keywords: Duloxetine, Osteoarthritis, Kurdistan Region
MeSH Terms: conditions — Osteoarthritis | interventions — Duloxetine Hydrochloride; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups, first group (case) will receive duloxetine tablet 30mg for two weeks then titrated up to duloxetine 30mg BID. Patients will be instructed to take the medication with meals.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine tablet (Active Comparator): Patient in the first group (case) will receive duloxetine tablet 30mg for two weeks then titrated up to duloxetine 30mg BID. Patients will be instructed to take the medication with meals for 13 weeks .
  Interventions: Drug: Duloxetine 30 MG; Drug: Nonsteroidal Antiinflammatory Drug
- NSAID(non steroidal anti inflammatory) (Active Comparator): patient in the second group will receive NSAID(non-steroidal anti inflammatory) drugs for 13 weeks
  Interventions: Drug: Duloxetine 30 MG; Drug: Nonsteroidal Antiinflammatory Drug

INTERVENTIONS:
Drug: Duloxetine 30 MG — patient in first group (case) will receive duloxetine tablet 30mg for two weeks then titrated up to duloxetine 30mg BID. Patients will be instructed to take the medication with meals. The for 13 weeks
  Other Names: Cymbalta
Drug: Nonsteroidal Antiinflammatory Drug — patient in this second group will receive NSAID for 3 weeks
  Other Names: NSAID

SUMMARY:
Osteoarthritis (OA) is the most common degenerative joint disease, affecting more than 25% of the population . Knee OA is an insidious disease related to structural changes in the joint over many years. Progressive articular damage results in a loss of the extracellular matrix of cartilage in addition to changes in subchondral bone.

Duloxetine, a selective serotonin, and norepinephrine reuptake inhibitor, it seems to be effective in treating neuropathic and chronic pain conditions.

DETAILED DESCRIPTION:
This will be a 13-week A randomized open labelled clinical trail in Iraqi Kurdistan Region, that will be designed to assess the efficacy of duloxetine tablet compared with other group (Nonsteroidal anti-inflammatory) drug on the reduction of pain caused by osteoarthritis of the knee.

Patients will be divided into two groups, first group (case) will receive duloxetine tablet 30mg for two weeks then titrated up to duloxetine 30mg BID. Patients will be instructed to take the medication with meals. Patients will be observed at visits (0) baseline then at second visits at 13 weeks then will be compared to control group that will receive NSAID (nonsteroidal anti-inflammatory drug) at baseline (0) visit then 2nd visits at 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. > 40years of age
2. both Genders
3. who will meet the American College of Rheumatology clinical and radiographic criteria for the diagnosis of osteoarthritis of the knee
4. with pain for ≥14days of each separate month for 3months before study entry, with a mean score ≥4 on the 24-h average pain score (0-10) using the average of daily ratings

Exclusion Criteria:

1. if they have diagnosed with inflammatory arthritis or an autoimmune disease
2. if they received invasive therapy in last 3 months (knee arthroscopy) or knee replacement at any time
3. patients with psychiatric disorders
4. Hypertension
5. Heart disease
6. patients on antipsychotics or anti-depressant -

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
twenty four hour 24-h average pain scores (short form) in patients with osteoarthritis knee pain | follow-up patients within two months
  it will report in patients' diaries based on the 11-point Likert scale (an ordinal scale with 0 indicating 'no pain', and 10 indicating 'worst pain imaginable')
(WOMAC) WESTERN ONTARIO AND MCMASTER OSTEOARTHITIS INDEX used for evaluation of pain in knee Osteoarthritis | follow-up patients within two months
  which involve three category about rating of pain(5 item) , stiffness(2item), physical function(17 item

SECONDARY OUTCOMES:
The other modality (clinical global improvement) | follow-up patients within two months
  will be used for severity of modality of pain and therapeutic response even side effect of drug

CONTACTS AND LOCATIONS:
Overall Officials: Aryan MF jalal, M.B.CH.B, Principal Investigator — Rheumatology , Hawler Medical University, Kurdistan Board for medical specialties; Niaz Albarzinji, MBCHB,DRMR, Study Director — Rheumatology, Hawler medical university/college of medicine
Locations (1):
- Rizgary and Cmc Hospital, Erbil, Iraq